CLINICAL TRIAL: NCT01422304
Title: A Randomized, Controlled, Parallel-group, Double-blind Trial of Sugammadex or Usual Care (Neostigmine or Spontaneous Recovery) for Reversal of Rocuronium- or Vecuronium-induced Neuromuscular Blockade in Patients Receiving Thromboprophylaxis and Undergoing Hip Fracture Surgery or Joint (Hip/Knee) Replacement (Protocol No. P07038)
Brief Title: Reversal of Neuromuscular Blockade With Sugammadex or Usual Care in Hip Fracture Surgery or Joint (Hip/Knee) Replacement (P07038)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P07038; 2011-001201-27 (EudraCT Number); MK-8616-059 (Other: Merck protocol number)
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Neuromuscular Blockade; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Blood Coagulation; Antithrombotic Agents
MeSH Terms: conditions — Thrombosis | interventions — Sugammadex; Neostigmine; Glycopyrrolate; Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex (Experimental): Prior to randomization, participants will be assigned to planned active reversal or planned spontaneous recovery by the anesthesiologist according to the recovery method the anesthesiologist would have chosen if the participant were not in the study. In this treatment arm, participants assigned to planned active reversal will receive sugammadex and placebo to neostigmine, and participants assigned to planned spontaneous recovery will receive sugammadex. Study drug will be administered after the last dose of rocuronium or vecuronium and after wound closure.
  Interventions: Drug: Sugammadex; Drug: Placebo to neostigmine
- Usual Care (Experimental): Prior to randomization, participants will be assigned to planned active reversal or planned spontaneous recovery by the anesthesiologist according to the recovery method the anesthesiologist would have chosen if the participant were not in the study. In this treatment arm, participants assigned to planned active reversal will receive neostigmine and placebo to sugammadex, and participants assigned to planned spontaneous recovery will receive placebo to sugammadex. Study drug will be administered after the last dose of rocuronium or vecuronium and after wound closure.
  Interventions: Drug: neostigmine and glycopyrrolate or atropine; Drug: Placebo to sugammadex

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 4 mg/kg intravenously
  Other Names: SCH 900616, MK-8616
  Arms: Sugammadex
Drug: neostigmine and glycopyrrolate or atropine — Neostigmine and glycopyrrolate or neostigmine and atropine administered intravenously per usual practice and per the product labels
  Arms: Usual Care
Drug: Placebo to neostigmine — Normal saline (NaCl 0.9%)
  Arms: Sugammadex
Drug: Placebo to sugammadex — Normal saline (NaCl 0.9%)
  Arms: Usual Care

SUMMARY:
This study will assess the effect of reversal of neuromuscular blockade with sugammadex compared with reversal according to usual care (neostigmine or spontaneous reversal) on the incidence of post-surgical bleeding events and on coagulation parameters in participants undergoing hip fracture surgery or joint (hip/knee) replacement surgery with neuromuscular blockage induced by rocuronium or vecuronium.

DETAILED DESCRIPTION:
Participants will be randomized to sugammadex or usual care in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Must be American Society of Anesthesiologists (ASA) Class 1, 2, or 3
* Must be scheduled for a hip fracture surgery or joint (hip or knee) replacement surgery under general anesthesia including the use of rocuronium or vecuronium for neuromuscular blockade
* Must be:

  * Currently receiving thromboprophylactic (anti-clotting) therapy with low molecular weight heparin (LMWH) or unfractionated heparin (UFH), or
  * Planned to initiate thromboprophylactic therapy with LMWH or UFH prior to or during surgery, or
  * Currently receiving ongoing thromboprophylactic therapy with a vitamin K antagonist that has been temporarily substituted with peri-operative LMWH or UFH, and/or
  * Currently receiving ongoing thromboprophylactic therapy with low-dose aspirin or other antiplatelet therapy
* Platelet count above the lower limit of normal range
* Appropriate candidate for rapid reversal of neuromuscular blockade
* Sexually active females must agree to use a medically accepted method of contraception through seven days after receiving protocol-specified medication

Exclusion Criteria:

* Anatomical malformations that may lead to difficult intubation
* Neuromuscular disorder that may affect neuromuscular blockade
* History of a coagulation disorder, bleeding diathesis, systemic lupus erythematosus or antiphospholipid syndrome
* History or evidence of active abnormal bleeding or blood clotting within 30 days prior to screening
* Significant hepatic dysfunction
* Severe renal insufficiency
* History or family history of malignant hyperthermia
* Hypersensitivity or hypersensitivity-like reaction to sugammadex, muscle relaxants, or other medications used during general anesthesia
* Planned intravenous administration of toremifene and/or fusidic acid within 24 hours before or within 24 hours after study medication
* Recent, severe trauma
* Body Mass Index (BMI) > 35
* Any contraindication to administration of sugammadex or neostigmine/glycopyrrolate (or neostigmine/atropine)
* Pregnant or intends to become pregnant between randomization and the Day 30 follow-up visit
* Breast-feeding
* Previously treated with sugammadex or participated in a sugammadex clinical trial
* Has an active hip/knee infection and is scheduled for revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2012-09-26 (Actual); Study Completion 2012-09-26 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rahe-Meyer N, Fennema H, Schulman S, Klimscha W, Przemeck M, Blobner M, Wulf H, Speek M, McCrary Sisk C, Williams-Herman D, Woo T, Szegedi A. Effect of reversal of neuromuscular blockade with sugammadex versus usual care on bleeding risk in a randomized study of surgical patients. Anesthesiology. 2014 Nov;121(5):969-77. doi: 10.1097/ALN.0000000000000424. PMID 25208233

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: For participants in this Arm assigned to planned active reversal of neuromuscular blockade: single intravenous (IV) administration of sugammadex 4 mg/kg and single IV administration of placebo (normal saline [NaCl 0.9%] to match volume of neostigmine/glycopyrrolate [or neostigmine/atropine] that would have been administered). For participants in this Arm assigned to planned spontaneous recovery from neuromuscular blockade: single IV administration of sugammadex 4 mg/kg.
- Usual Care: For participants in this Arm assigned to planned active reversal of neuromuscular blockade: single IV administration of neostigmine (up to a maximum dose of 5 mg) with glycopyrrolate or atropine and single IV administration of placebo (normal saline [NaCl 0.9%] to match volume of sugammadex that would have been administered). For participants in this Arm assigned to planned spontaneous recovery from neuromuscular blockade: single IV administration of placebo (normal saline [NaCl 0.9%] to match volume of sugammadex that would have been administered).
Period: Overall Study
Arm/Group | Sugammadex | Usual Care
Started | 598 (Randomized) | 600 (Randomized)
Treated | 595 | 589 (1 given sugammadex; thus All Participants as Treated (APaT) Ns are 596 Sugammadex, 588 Usual Care)
Completed | 574 | 563
Not Completed | 24 | 37
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 14 | 20
Not completed — Never Entered Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Did Not Meet Protocol Eligibility | 0 | 2
Not completed — Not Treated | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Usual Care | Total
Number analyzed (Participants) | 596 | 588 | 1184
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (12.0) | 66.6 (11.3) | 66.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 340 | 666
  Male | 270 | 248 | 518
Activated Partial Thromboplastin Time (aPTT) [Mean (Standard Deviation); unit: seconds] — n=556, 535, 1091 for Sugammadex, Usual Care and Total, respectively
  seconds | 31.14 (4.38) | 31.01 (4.14) | 31.08 (4.26)
Prothrombin Time (International Normalized Ratio) (PT[INR]) [Mean (Standard Deviation); unit: ratio] — n=557, 535, 1092 for Sugammadex, Usual Care and Total, respectively
  ratio | 1.121 (0.159) | 1.114 (0.132) | 1.117 (0.147)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adjudicated Events of Bleeding (Major or Non-major) With Onset Within 24 Hours After Study Drug Administration
Description: Post-treatment events of bleeding were evaluated by a medically-qualified, blinded member of the surgical team (Blinded Safety Assessor), in consultation with the surgeon, to determine if an event was a "suspected, unanticipated adverse event of bleeding" (SUAEB). A SUAEB is an event of bleeding outside the usual boundaries of expectations for a participant (e.g., in amount of blood lost, prolonged duration of bleeding, or other factors) considering the type of procedure as well as participant's specific surgical experience and underlying risk of bleeding. In addition, blinded review of clinical and laboratory databases was performed to identify any event potentially consistent with a SUAEB; these were reviewed by the Blinded Safety Assessor, who determined if any was a SUAEB. All SUAEBs were evaluated by a blinded external Adjudication Committee, which classified each as either: 1) a major bleeding event, 2) a non-major bleeding event, or 3) not an unanticipated event of bleeding.
Time Frame: Up to 24 hours post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 17 | 24
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Cochran-Mantel-Haenszel method was stratified for renal function (estimated creatinine clearance < or ≥ 60 mL/min) and prophylactic antithrombotic therapy (including low molecular weight heparin [LMWH], including unfractionated heparin [UFH], or not including either LMWH or UFH); Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.38 to 1.29] — Relative risk is Sugammadex versus Usual Care

2. Secondary Outcome: Percent Change From Baseline in Activated Partial Thromboplastin Time (aPTT) at 10 and 60 Minutes Post Study Drug Administration
Description: Change from baseline in aPTT is identified in study protocol as the Key Secondary Outcome Measure. Blood samples for determination of aPTT values were obtained at baseline and at 10 and 60 minutes after study drug administration. aPTT is a performance indicator measuring the efficacy of the intrinsic and common blood coagulation (blood clotting) pathways. Higher values of aPTT indicate a reduction in the clotting tendency of blood.
Time Frame: Baseline, 10 and 60 minutes post study drug administration
Population: Participants in APaT population who had baseline and at least one post baseline aPTT measurement within defined assessment window (10 or 60 minutes post study drug).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 556 | 535
percent change
  10 minutes (Sugammadex n=525, Usual Care n=507) | 6.0 (22.4) [3.4 to 5.9] | -0.1 (13.6) [-2.0 to 0.4]
  60 minutes (Sugammadex n=523, Usual Care n=505) | 0.4 (29.1) | -1.2 (22.7)
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Model was restricted to have no difference between treatment groups for baseline assessment, and was adjusted for center, usual care group (active reversal or spontaneous recovery), renal function (estimated creatinine clearance < or ≥ 60 mL/min), prophylactic antithrombotic therapy (including LMWH, including UFH, or not including either LMWH or UFH), type of hip/knee surgical procedure, and the interaction of time by treatment; Test type: Superiority or Other; Constrained Longitudinal Data Analysis; Model included those in APaT population with any baseline or post baseline aPTT value in 10 or 60 minute window (Sugammadex, Usual Care N=567, 548); Geometric Mean Ratio (GMR) (%) = 5.5, 95% CI 2-sided [3.7 to 7.3] — Estimate of difference in Sugammadex versus Usual Care change from baseline at 10 minutes post dose calculated with log of aPTT values as dependent variable. Results transformed back to GMR of respective changes (expressed as %, = [GMR - 1]*100)
Statistical Analysis 2: Comparison: Sugammadex vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Constrained Longitudinal Data Analysis; [statistical method as in outcome 2, analysis 1]; GMR (%) = 0.9, 95% CI [-0.9 to 2.8] — Estimate of difference in Sugammadex versus Usual Care change from baseline at 60 minutes post dose calculated with log of aPTT values as dependent variable. Results transformed back to GMR of respective changes (expressed as %, = [GMR - 1]*100)

3. Secondary Outcome: Percent Change From Baseline in Prothrombin Time (International Normalized Ratio) (PT[INR]) at 10 and 60 Minutes Post Study Drug Administration
Description: Change from baseline in PT(INR) is identified in study protocol as an Other Secondary Outcome Measure. Blood samples for determination of PT(INR) values were obtained at baseline and at 10 and 60 minutes after study drug administration. PT(INR) is a performance indicator measuring the efficacy of the extrinsic and common blood coagulation (blood clotting) pathways. The INR is the ratio of a participant's prothrombin time to a normal (control) sample, raised to the power of the International Sensitivity Index (ISI) value for the analytical system used (INR = [PT-Test/PT-Normal]^ISI). Higher values of PT(INR) indicate a reduction in the clotting tendency of blood.
Time Frame: Baseline, 10 and 60 minutes post study drug administration
Population: Participants in APaT population who had baseline and at least one post baseline PT(INR) measurement within defined assessment window (10 or 60 minutes post study drug).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 557 | 535
percent change
  10 minutes (Sugammadex n=526, Usual Care n=507) | 8.0 (63.4) | 2.5 (14.3)
  60 minutes (Sugammadex n=524, Usual Care n=505) | 8.9 (79.8) | 3.4 (23.2)
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Constrained Longitudinal Data Analysis; Model included those in APaT population with any baseline or post baseline PT(INR) value in 10 or 60 minute window (Sugammadex, Usual Care N=567, 548); GMR (%) = 3.0, 95% CI 2-sided [1.3 to 4.7] — Estimate of difference in Sugammadex versus Usual Care change from baseline at 10 minutes post dose calculated with log of PT(INR) values as dependent variable. Results transformed back to GMR of respective changes (expressed as %, = [GMR - 1]*100)
Statistical Analysis 2: Comparison: Sugammadex vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Constrained Longitudinal Data Analysis; [statistical method as in outcome 3, analysis 1]; GMR (%) = 0.9, 95% CI 2-sided [-1.0 to 2.9] — Estimate of difference in Sugammadex versus Usual Care change from baseline at 60 minutes post dose calculated with log of PT(INR) values as dependent variable. Results transformed back to GMR of respective changes (expressed as %, = [GMR - 1]*100)

4. Secondary Outcome: Number of Participants With One or More Adjudicated Events of Bleeding (Major or Non-major) With Onset Within 14 Days After Study Drug Administration
Description: This Measure is identified in study protocol as an Other Secondary Outcome Measure. Post-treatment events of bleeding were evaluated by a medically-qualified, blinded member of the surgical team (Blinded Safety Assessor), in consultation with the surgeon, to determine if an event was a "suspected, unanticipated adverse event of bleeding" (SUAEB). A SUAEB is an event of bleeding outside the usual boundaries of expectations for a participant considering the type of procedure as well as participant's specific surgical experience and underlying risk of bleeding. In addition, blinded review of clinical and laboratory databases was performed to identify any event potentially consistent with a SUAEB; these were reviewed by the Blinded Safety Assessor, who determined if any was a SUAEB. All SUAEBs were evaluated by a blinded external Adjudication Committee, which classified each as either: 1) a major bleeding event, 2) a non-major bleeding event, or 3) not an unanticipated event of bleeding.
Time Frame: Up to 14 days post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 24 | 27
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = -0.6, 95% CI 2-sided [-3.0 to 1.8] — Risk difference (%) = Sugammadex incidence - Usual Care incidence

5. Secondary Outcome: Number of Participants With One or More Adjudicated Major Events of Bleeding With Onset Within 24 Hours After Study Drug Administration
Description: This Measure is identified in study protocol as an Other Secondary Outcome Measure. All SUAEB were evaluated by a blinded external Adjudication Committee. Major bleeding event (MBE) = one or more of the following: 1) Fatal bleeding; 2) Bleeding that is symptomatic and occurs in critical area/organ, in a non-operated joint, or is intramuscular with compartment syndrome; 3) Extrasurgical site bleeding causing a fall in hemoglobin (Hgb) level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red blood cells (RBCs), occurring within 24 hours of the bleeding; 4) Surgical site bleeding requiring second intervention, or bleeding at operated joint that interferes with rehabilitation; or 5) Surgical site bleeding that is unexpected/prolonged and/or causes hemodynamic instability, with fall in Hgb level of at least 20 g/L (1.24 mmol/L) or transfusion of at least two units of whole blood or RBCs, occurring within 24 hours of the bleeding.
Time Frame: Up to 24 hours post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 12 | 20
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = -1.4, 95% CI 2-sided [-3.4 to 0.5] — Risk difference (%) = Sugammadex incidence - Usual Care incidence

6. Secondary Outcome: Number of Participants With One or More Adjudicated Major Events of Bleeding With Onset Within 14 Days After Study Drug Administration
Description: This Measure is identified in study protocol as an Other Secondary Outcome Measure. All SUAEB were evaluated by a blinded external Adjudication Committee. MBE = one or more of the following: 1) Fatal bleeding; 2) Bleeding that is symptomatic and occurs in critical area/organ, in a non-operated joint, or is intramuscular with compartment syndrome; 3) Extrasurgical site bleeding causing a fall in Hgb level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or RBCs, occurring within 24 hours of the bleeding; 4) Surgical site bleeding requiring second intervention, or bleeding at operated joint that interferes with rehabilitation; or 5) Surgical site bleeding that is unexpected/prolonged and/or causes hemodynamic instability, with fall in Hgb level of at least 20 g/L (1.24 mmol/L) or transfusion of at least two units of whole blood or RBCs, occurring within 24 hours of the bleeding.
Time Frame: Up to 14 days post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 18 | 23
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = -0.9, 95% CI 2-sided [-3.1 to 1.2] — Risk difference (%) = Sugammadex incidence - Usual Care incidence

7. Secondary Outcome: Number of Participants With One or More Adjudicated Venous Thromboembolic (VTE) Events With Onset Within 14 Days After Study Drug Administration
Description: This Measure is identified in study protocol as an Other Secondary Outcome Measure. Suspected symptomatic VTE events were evaluated by a blinded external Adjudication Committee. The confirmation of a VTE event was based on determination of a clinically meaningful venous thrombosis (e.g., pulmonary embolism or deep vein thrombosis).
Time Frame: Up to 14 days post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 5 | 3
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = 0.3, 95% CI 2-sided [-0.7 to 1.5] — Risk difference (%) = Sugammadex incidence - Usual Care incidence

8. Secondary Outcome: Number of Participants With One or More Adjudicated Events of Anaphylaxis With Onset Within 14 Days After Study Drug Administration
Description: This Measure is identified in study protocol as an Other Secondary Outcome Measure. Anaphylaxis is a serious allergic reaction that is rapid in onset and may cause death. Adverse events suggestive of hypersensitivity which met defined criteria (e.g., serious event) and/or suspected events of anaphylaxis were evaluated by a blinded external Adjudication Committee to determine whether such events met either of the following two criteria for anaphylaxis (Sampson et al. J Allergy Clin Immunol 2006;117:391-7) - 1. Acute onset of an illness with involvement of the skin, mucosal tissue or both, and at least one of the following: a) respiratory compromise, b) reduced blood pressure (BP) or associated symptoms of end-organ dysfunction. 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that participant: a) involvement of the skin-mucosal tissue, b) respiratory compromise, c) reduced BP or associated symptoms, d) persistent gastrointestinal symptoms.
Time Frame: Up to 14 days post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 0 | 0

9. Other Pre Specified Outcome: Postoperative Drainage Volume Within 24 Hours After Study Drug Administration
Description: The total volume of postoperative drainage from the surgical site over the 24 hours after study drug administration was recorded.
Time Frame: Up to 24 hours post study drug administration
Population: APaT population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
mL | 464 (367.5) | 476 (375.3)
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Generalized Linear Model was adjusted for strata (renal function and use of prophylactic antithrombotic therapy) and investigational site; Test type: Superiority or Other; Generalized Linear Model; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-45.0 to 30.5] — Difference is Sugammadex versus Usual Care. A negative value indicates that the average adjusted drainage volume was lower in the sugammadex treatment group

10. Other Pre Specified Outcome: Number of Participants Requiring Any Postoperative Transfusion
Description: The number of participants who received a transfusion unit (e.g., whole blood, packed RBCs, cell saver RBCs, fresh frozen plasma, platelets) that started after study drug administration and within 120 hours after study drug administration (or within 48 hours after any previous [i.e., predose] transfusion for participants who had received a previous transfusion) was determined.
Time Frame: From end of study drug administration through approximately 120 hours after study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 221 | 227
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Miettinen and Nurminen Method was adjusted for strata (renal function and use of prophylactic antithrombotic therapy) and investigational site; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = -2.7, 95% CI 2-sided [-7.4 to 2.0] — Risk difference (%) = Sugammadex incidence - Usual Care incidence, adjusted for strata and investigational site

11. Other Pre Specified Outcome: Total Transfusion Volume in Participants Who Required Postoperative Transfusion
Description: Among participants who received a transfusion unit (e.g., whole blood, packed RBCs, cell saver RBCs, fresh frozen plasma, platelets) that started after study drug administration and within 120 hours after study drug administration (or within 48 hours after any previous [i.e., predose] transfusion for participants who had received a previous transfusion), the total volume of blood transfused post study drug was calculated. The volume of blood transfused post study drug (using linear interpolation when transfusions were ongoing at the time of study drug administration) was converted to grams of Hgb transfused, using RBC concentration information received from the investigators. The sum of Hgb transfused was standardized to "normal" volume Hgb in homologous whole blood, using 20 g/dL Hgb for calculation of the standardized volume.
Time Frame: From end of study drug administration through approximately 120 hours after study drug administration
Population: Participants in APaT population who received a transfusion unit that started after study drug administration and within 120 hours after study drug administration (or within 48 hours after any previous [i.e., predose] transfusion for participants who had received a previous transfusion)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 221 | 227
mL | 335 (74) | 345 (84.5)
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Generalized Linear Model was applied to transfusion volume transformed to the log-scale, adjusted for strata (renal function and use of prophylactic antithrombotic therapy) and investigational site. Result and 95% Confidence Interval was transformed back to the original scale; Test type: Superiority or Other; Generalized Linear Model; GMR = 1.10, 95% CI 2-sided [0.98 to 1.24] — GMR is Sugammadex versus Usual Care

12. Other Pre Specified Outcome: Postoperative Changes in Hgb Concentrations Using the Bleeding Index
Description: The Bleeding Index was used to describe postoperative changes in Hgb concentrations at Visit 3. Bleeding Index = Hgb level at Visit 3 - Hgb level at baseline, adjusted for the amount of RBCs transfused. Missing baseline Hgb values were imputed using the overall mean Hgb value at baseline.
Time Frame: Baseline and Visit 3 (24-48 hours post study drug administration)
Population: APaT population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
g/L | -15.7 (15.7) | -17.4 (17.1)
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Generalized Linear Model was adjusted for strata (renal function and use of prophylactic antithrombotic therapy), investigational site and baseline hemoglobin value; Test type: Superiority or Other; Generalized Linear Model; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.4 to 3.1] — Difference is Sugammadex versus Usual Care. A positive value indicates that the average adjusted reduction in Hgb at Visit 3 (bleeding index) was lower in the sugammadex treatment group

13. Other Pre Specified Outcome: Number of Participants With One or More Postoperative Anemia Adverse Events With Onset Within 72 Hours After Study Drug Administration
Description: This measure is the incidence of postoperative anaemia with an onset within 72 hours after study drug administration. A participant is included in the count for this measure if an adverse event with any of the following event terms occurred in the participant with onset within the defined time frame: postoperative anaemia, anaemia, haemorrhagic anaemia, haemoglobin decreased or haemoglobin S decreased.
Time Frame: Up to 72 hours post study drug administration
Population: APaT population
Measure: Number; unit: participants
Arm/Group | Sugammadex | Usual Care
Number analyzed (Participants) | 596 | 588
participants | 124 | 132
Statistical Analysis 1: Comparison: Sugammadex vs Usual Care; Test type: Superiority or Other; Miettinen and Nurminen; Risk Difference (%) = -1.6, 95% CI 2-sided [-6.3 to 3.1] — Risk difference (%) = Sugammadex incidence - Usual Care incidence

ADVERSE EVENTS:
Time Frame: Up to 14 days post study drug administration
Description: Adverse event tables include participants in APaT population
Arm/Group | Sugammadex | Usual Care
Serious Adverse Events (participants affected / at risk) | 39/596 | 40/588
Other Adverse Events (participants affected / at risk) | 491/596 | 499/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=596) | Usual Care (N=588)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Device breakage (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 4 (4)
Pain (General disorders) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femoral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Supportive care (Surgical and medical procedures) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=596) | Usual Care (N=588)
Anaemia (Blood and lymphatic system disorders) | 72 (75) | 74 (74)
Constipation (Gastrointestinal disorders) | 128 (129) | 146 (148)
Nausea (Gastrointestinal disorders) | 124 (138) | 139 (154)
Vomiting (Gastrointestinal disorders) | 64 (67) | 70 (74)
Oedema peripheral (General disorders) | 53 (55) | 47 (50)
Pain (General disorders) | 91 (112) | 101 (124)
Anaemia postoperative (Injury, poisoning and procedural complications) | 63 (64) | 65 (66)
Procedural pain (Injury, poisoning and procedural complications) | 203 (224) | 234 (259)
Hypokalaemia (Metabolism and nutrition disorders) | 33 (33) | 45 (47)
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 (84) | 40 (60)
Insomnia (Psychiatric disorders) | 50 (50) | 54 (55)
Sleep disorder (Psychiatric disorders) | 87 (90) | 84 (86)
Erythema (Skin and subcutaneous tissue disorders) | 26 (31) | 32 (38)
Haematoma (Vascular disorders) | 59 (61) | 53 (54)
Hypotension (Vascular disorders) | 27 (28) | 37 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Initial public presentation of the Investigator's results will occur only together with the other sites unless permission is obtained from Sponsor. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. In case of disagreement concerning appropriateness of materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues, prior to submission for publication/presentation.